CLINICAL TRIAL: NCT05065528
Title: A Randomized Trial Evaluating the Efficacy of Oral Magnesium in Symptomatic Reduction of Acute Concussion in Adolescents
Brief Title: Mag Con: Efficacy of Oral Mag. in Acute Concussion in Adolescents
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Did not recruit any participants
Sponsor: Corewell Health South (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: EGME#01-2021
Record Dates: First submitted 2021-09-23; First posted 2021-10-04 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Concussion, Mild; Traumatic Brain Injury, Mild
MeSH Terms: conditions — Brain Concussion | interventions — Magnesium

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Placebo Comparator): placebo pill twice daily for 3 days ondansetron 4mg twice daily for 3 days acetaminophen 500mg twice daily for 3 days
  Interventions: Drug: Placebo
- Intervention (Experimental): Magnesium 500mg twice daily for 3 days ondansetron 4mg twice daily for 3 days acetaminophen 500mg twice daily for 3 days
  Interventions: Dietary Supplement: Magnesium

INTERVENTIONS:
Dietary Supplement: Magnesium — Will receive symptomatic care (ondansetron 4mg and acetaminophen 500 mg each twice daily) along with 400 mg supplemental magnesium twice daily for 3 days
  Arms: Intervention
Drug: Placebo — Will receive symptomatic care (ondansetron 4mg and acetaminophen 500 mg each twice daily) along with placebo pill
  Arms: Control

SUMMARY:
This randomized trial will compare the clinical efficacy of adding oral magnesium oxide to acetaminophen and ondansetron in the treatment of adolescents presenting within 48 hours of a mild traumatic brain injury using the Post-Concussion Symptom Severity Score Index.

DETAILED DESCRIPTION:
This randomized trial will compare the clinical efficacy of oral magnesium oxide, acetaminophen and ondansetron, to that of PO acetaminophen and ondansetron in the treatment of adolescents presenting within 48 hours of a mild traumatic brain injury. Our primary endpoint will be to evaluate if magnesium has an impact on patient's Post-Concussion Symptom Severity Score Index. This will be evaluated both at the initial presentation in-person and then at 24, 48, and 72 hours via phone

ELIGIBILITY:
Inclusion Criteria:

* age 12 to 18 years;
* presenting chief complaint of headache, head injury, or concussion within the first 48 hours of injury;
* GCS > 13 on arrival

Exclusion Criteria:

* age < 12 years or > 18 years;
* inability to provide informed consent;
* vomiting > 2 episodes following injury;
* physical or mental disability hindering adequate response to assessment of symptoms;
* hemodynamic instability/medical condition requiring further acute life-saving medical intervention;
* known brain mass, intracranial hemorrhage, skull fracture;
* known contraindications/allergy to magnesium, ondansetron, or acetaminophen
* pregnant patients

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Post-Concussion Symptom Severity Score | 48, 72 hours
  The Post-Concussion Symptom Severity Score is a validated score measuring concussion symptoms and intensity. It measures 22 symptoms on a scale from 0 to 6. The score therefore ranges from 0 (no symptoms) through 132 (maximal symptoms). These will be evaluated at baseline as well as 48 and 72 hours from treatment. Means for each group will be calculated and compared

SECONDARY OUTCOMES:
adverse effect related to medication administration | 48, 72 hours
  proportion of patients in each group who have developed of adverse effects related to medication administration
return to baseline | 48, 72 hours
  proportion of patients in each group who have experienced symptom resolution

CONTACTS AND LOCATIONS:
Overall Officials: Chris Trigger, DO, Principal Investigator — Corewell Health South
Locations (1):
- Spectrum Health Lakeland, Saint Joseph, Michigan, United States

IPD SHARING:
Plan to Share IPD: No